## Confidential

Page 1

mPATH Staff Survey - Consent & Contact Information

IMPLEMENTATION OF MPATH™

David P. Miller, MD, MS, Principal Investigator

Study Information Sheet for Staff Surveys

You are being asked to participate in a survey study. Your participation is voluntary. There is no penalty for choosing not to participate. You are being asked to take part in this study because you work at a clinic that is using the mPATH

iPad app. About 300 people from 30 primary care clinics will participate in this study.

WHY IS THIS STUDY BEING DONE?

We are conducting this study because we want to learn the best way to implement a new iPad program in clinical practice.

WHAT IS INVOLVED?

You will be asked to complete up to three surveys over one year. Each survey takes less than 10 minutes to complete.

WHAT ARE THE RISKS, COSTS, AND BENEFITS OF PARTICIPATING IN THE STUDY?

The risk of harm or discomfort that may happen as a result of taking part in this research study is not expected to be more than in daily life. There is no cost to participate. You are not expected to receive any direct benefit from takingpart in this research study. We hope the information learned from this study will benefit clinics in the future.

WILL I BE PAID?

You will receive a \$10 gift card for each survey you complete as a token of thanks for your time.

Dr. David Miller and Dr. Ajay Dharod are the developers of the mPATH™ application. Dr. Miller, Dr. Dharod, and Wake

Forest University Health Sciences have an ownership interest in the application and may financially benefit from futures sales of the application related to this study. There are no plans to provide you with financial compensationor for you to share in any profits if this should occur.

WHAT ABOUT CONFIDENTIALITY?

To keep your information confidential, we will assign you a unique study identifier. Only your anonymous study identifier will be stored with your survey answers. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe. We will not include your name in any report we might publish.

## WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

If you have questions about the study, please ask them now.

If you later have questions, you may contact the study investigator, Dr. David Miller at 336-713-4156. The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB at (336) 716-4542.

## WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

You may choose not to take part or you may leave the study at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff. The investigators also have the right to stop your participation in the study at any time. Information about you may be removed from the study data and could be used for future research or shared with other researchers without additional consent from you.

By continuing, I agree to take part in this study. I authorize the use and disclosure of my information as described in this consent and authorization form. I have had a chance to ask questions about being in this study and have those questions answered. By taking part in the study, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

| Last Name |
|------------------------------------------------------|
| Wake Health Email Address |
| (We may send you up to two additional surveys) |
| Clinic Reynolda Family Medicine |
| Bermuda Run Family Medicine |
| Conover Family Medicine |
| Catawba Internal Medicine |
| Westchester Internal Medicine |
| High Point Premier Internal Medicine |
| Archdale Family Medicine |
| Adams Farm Family Medicine |
| Please click "Submit" to move on to the next survey. |

First Name